CLINICAL TRIAL: NCT05656703
Title: Monitoring of Anesthesia Depth Reduces the Incidence of Postoperative Delirium and Preserves Memory Abilities Better in the High Risk Elderly
Brief Title: Anesthesia Depth Increases Delirium Incidence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Thomas Frietsch, Associate Professor, Heidelberg University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2013-627N-MA
Record Dates: First submitted 2022-05-12; First posted 2022-12-19 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: Delirium; Anesthesia Awareness
Keywords: bispectral index monitoring; anesthesia depth
MeSH Terms: conditions — Delirium; Intraoperative Awareness | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Randomised-controlled, double blind study, monocentric
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: group blinding for all of the above except for staff anesthesiologist of the light anesthesia group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bis Guided light anesthesia (Experimental): Patients are monitored by bispectral index and held under light anesthesia (BIS level 45 to 60)
  Interventions: Device: BIS guidance of anesthesia
- Standard of Care (Placebo Comparator): Patients receive standard of care anesthesia, BIS monitor was covered with a blind
  Interventions: Other: Standard of Care

INTERVENTIONS:
Device: BIS guidance of anesthesia — Anesthesia is to be directed to a specific (light) level by the dosage of administered hypnotics and analgesics
  Arms: Bis Guided light anesthesia
Other: Standard of Care — Anesthesia is administered as usual
  Arms: Standard of Care

SUMMARY:
This study aimed to determine whether targeting bispectral index (BIS) readings of 55 (light anaesthesia) was associated with a lower incidence of delirium, dementia (POD), POCD and mortality but higher rates of awareness and complications than a standard of care anaesthesia blinded to depth monitoring.

DETAILED DESCRIPTION:
Design: Randomised-controlled, double blind study, monocentric Setting: Level 2 medical center, major surgery (non cardiac) Ethics: Ethical approval for this study (Ethikkommission II der Ruprecht-Karls-Universität Heidelberg 2013-627N-MA) was provided by the Ethical Committee II University Medicine Mannheim, University of Heidelberg, Germany (Chairperson Prof W. Striebel) on Mai 12th 2008.

Patients: n=130, aged > 70y Intervention: Light anesthesia (BIS 55 +/-5) vs. Standard of Care (BIS- blinded) Main outcome measures: Incidence of awareness, delirium, postoperative cognitive deficit (POCD), dementia (POD), memory (MAT with a computerized score for verbal working&short term, figural working&short term memories and well as attention level) Second aims: mortality, complications

ELIGIBILITY:
Inclusion Criteria:

* scheduled for major surgery above 60 min duration
* informed consent

Exclusion Criteria:

* emergency surgery with large blood loss and/or preoperative cardiovascular instability, scheduled regional or neuraxial anesthesia, language barriers with the unability to understand a German audio tape, unability or unwillingness to consent,hearing disabilities

Ages: 70 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 130 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
postoperative delirium by NUDESC | 6 to 24 months
  in the hospital with NUDESC Score
postoperative dementia and cognitive deficit By MMSE and MAT Test | 6 to 24 months
  in the hospital by MMSE and MAT (automated computerized test), after discharge by a standardized questionnaire
awareness, memory function | 1 to 3 days postoperative
  implicit and explicit memory for intraoperative wakefulness and memory functions in general as changing conditions due to anesthesia

SECONDARY OUTCOMES:
mortality and morbidity | 6 to 24 months
  death rate (in hospital and longterm mortality (death/month)) and complication rate (in hospital and longterm morbidity (complications/month))

CONTACTS AND LOCATIONS:
Locations (1):
- Clinic of Anesthesiology and Critical Care Medicine, Faculty of Clinical Medicine MAnnheim, University of Heidelberg, Germany, Mannheim, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No